CLINICAL TRIAL: NCT00368290
Title: Modafinil Treatment for Cocaine Dependence and HIV-High Risk Behavior
Brief Title: Modafinil Treatment for Cocaine Dependence and HIV High-Risk Behavior
Acronym: MOD6
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyle Kampman (Other)
Responsible Party: Sponsor-Investigator, Kyle Kampman, Sponsor-Investigator, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 804537
Record Dates: First submitted 2006-08-22; First posted 2006-08-24 (Estimated); Results first posted 2014-01-29 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-02

CONDITIONS: Cocaine Dependence
Keywords: cocaine dependence; hiv prevention
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Modafinil; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): modafinil plus CBT
  Interventions: Drug: Modafinil; Behavioral: Cognitive Behavioral Therapy (CBT)
- 2 (Placebo Comparator): placebo plus CBT
  Interventions: Drug: placebo; Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Drug: Modafinil — 300mg a day for 8 weeks
  Other Names: Provigil
  Arms: 1
Drug: placebo — placebo pills for 8 weeks
  Arms: 2
Behavioral: Cognitive Behavioral Therapy (CBT) — Weekly cognitive behavioral therapy sessions for a period of 8 weeks.

SUMMARY:
The purpose of study is to determine if modafinil promotes cocaine abstinence and reduces high risk behavior in cocaine dependent subjects.

DETAILED DESCRIPTION:
The purpose of study is to determine if modafinil promotes cocaine abstinence and reduces HRB in cocaine dependent subjects. Modafinil (300 mg/day) or placebo will be administered in an 8-week double-blind trial to patients meeting diagnostic criteria for cocaine dependence in conjunction with Cognitive Behavioral Therapy (CBT).

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 60 years;
2. Current DSM-IV diagnosis of cocaine dependence;
3. Using cocaine at least 8 days in a consecutive 30 day period over the 60 day period immediately preceding study entry (If subject was receiving inpatient substance abuse treatment within 30 days prior to screening, subject must have been using cocaine at least 8 days in a consecutive 30 day period over the 60 day period immediately preceding admission to inpatient treatment); 4.)Having a negative urine toxicology (BE) test during screening (no less than 5 days prior to randomization) and a negative urine toxicology (BE) test on the day of randomization. Repeat testing allowed until required negative BE results are obtained;
4. Able to provide written informed consent and to comply with all study procedures;
5. Women must be surgically sterile, at least two years postmenopausal, or, if of childbearing potential, be using a medically accepted method of birth control and agree to continue use of this method for at least 30 days after the last dose of study drug (i.e. barrier method with spermicide, steroidal contraceptive [oral and implanted, including Depo-Provera, contraceptives must be used in conjunction with a barrier method], or intrauterine device [IUD]).

Exclusion Criteria:

1. Currently dependent on any substance other than cocaine or nicotine;
2. Current Neurological or psychiatric disorders, such as psychosis, bipolar illness, organic brain disease, dementia, or any diseases that require psychotropic medications;
3. Serious medical illnesses, including but not limited to; uncontrolled hypertension, significant heart disease (including a history of myocardial infarction, angina, mitral valve prolapse, left ventricular hypertrophy, palpitations, and arrhythmia), hepatic disease, renal disease, or any serious, potentially life-threatening or progressive medical illness that may compromise patient safety or study conduct;
4. Received a drug with known potential for toxicity to a major organ system within the month prior to entering treatment including, but not limited to: chemotherapeutic agents for neoplastic disease (i.e. methotrexate, vincristine, vinblastine, fluorouracil), agents used for parasitic infections, isoniazid, chlorambucil, dactinomycin, chloramphenicol, immunosuppressive and cytotoxic agents (i.e. cyclosporine, tacrolimus), indomethacin, protease inhibitors, amphotericin B, cephalosporins, aminoglycosides, interferon, and sulfonamides;
5. Clinically significant abnormal laboratory values (see Appendix A);
6. Has any disease of the gastrointestinal system, liver, or kidneys which could result in altered metabolism or excretion of the study medication (history of major gastrointestinal tract surgery, gastrectomy, gastrostomy, bowel resection, etc.) or history of chronic gastrointestinal disorders (ulcerative colitis, regional enteritis, or gastrointestinal bleeding);
7. Known hypersensitivity or allergy to modafinil, or receiving chronic therapy with any medication that could interact adversely with modafinil, including propranolol, phenytoin, warfarin and diazepam;
8. Took monoamine oxidase inhibitors (MAOI) within 30 days prior to randomization;
9. Taking or has taken an investigational drug within 60 days prior to randomization;
10. If female and of child-bearing capacity, tests positive on a urine pregnancy test, is lactating, has had three or more days of amenorrhea beyond expected menses at the time of the first dose of study medication, is contemplating pregnancy in the next 6 months, or is not using an effective contraceptive method;
11. Received therapy with any opiate-substitute (methadone, LAAM, buprenorphine) within 60 days of study enrollment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2006-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle M Kampman, M.D., Principal Investigator — University of Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Modafinil: modafinil plus CBT
  Modafinil: 300mg a day for 8 weeks
  Cognitive Behavioral Therapy (CBT): Weekly cognitive behavioral therapy sessions for a period of 8 weeks.
- Placebo: placebo plus CBT
  placebo: placebo pills for 8 weeks
  Cognitive Behavioral Therapy (CBT): Weekly cognitive behavioral therapy sessions for a period of 8 weeks.
Period: Overall Study
Arm/Group | Modafinil | Placebo
Started | 47 | 47
Completed | 34 | 37
Not Completed | 13 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modafinil | Placebo | Total
Number analyzed (Participants) | 47 | 47 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 47 | 94
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 38 | 39 | 77
Region of Enrollment [Number; unit: participants]
  United States | 47 | 47 | 94

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Reporting no Cocaine Craving
Description: Percent of participants reporting no cocaine craving based on Brief Substance Craving Scale (BSCS) - a 4 point likert scale.
Time Frame: 8 weeks
Measure: Number; unit: Percent of participants
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 47 | 47
Percent of participants | 64 | 41

2. Primary Outcome: Cocaine Use as Measured by Urine Drug Screen
Description: The primary outcome measure was cocaine use measured by self-report, and confirmed by twice weekly urine drug screens. The percentage of participants shows the percentage who were abstinent from cocaine during the last 3 weeks of the trial.
Time Frame: 8 weeks
Measure: Number; unit: Percentage of Participants
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 47 | 47
Percentage of Participants | 23 | 9

ADVERSE EVENTS:
Arm/Group | Modafinil | Placebo
Serious Adverse Events (participants affected / at risk) | 6/47 | 9/47
Other Adverse Events (participants affected / at risk) | 23/47 | 12/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modafinil (N=47) | Placebo (N=47)
Loss of Conciousness (General disorders) | 1 (1) | 0 (0) — Subject was driving and reportedly lost consciousness, causing his car to hit the side of a house. The expected charges are driving under the influence and malicious mischief with a motor vehicle.
Exacerbation of Cocaine Dependence (General disorders) | 3 (4) | 5 (5) — Subject's cocaine dependence let subject to enter an inpatient program.
Hospitalization for Depression (Psychiatric disorders) | 1 (1) | 2 (2) — Subject entered psychiatric treatment facility
Hospitalization for Asthama (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) — Subject hospitalized for worsening asthma symptoms
Hospitalization for eye injury (Eye disorders) | 0 (0) | 1 (1) — Subject was hospitalized for eye surgery
Infection in laceration on right hand (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Modafinil (N=47) | Placebo (N=47)
Headache (General disorders) | 6 | 7
Insomnia (General disorders) | 10 | 3
Anxiety (Psychiatric disorders) | 7 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No